CLINICAL TRIAL: NCT06404151
Title: Comparison of Oxygen Reserve Index and Regional Cerebral Oxygen Saturation in Determining Hypoxia in Obese Patients
Brief Title: Comparison of Oxygen Reserve Index and Regional Cerebral Oxygen Saturation Indetermining Hypoxia in Obese Patients
Status: Recruiting | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gülten Arslan, assos prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2023/514/246/17
Record Dates: First submitted 2024-02-28; First posted 2024-05-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Oxygen Deficiency
Keywords: Oxygen reserve index,; Preoxygenation; Cerebral Oxygen Saturation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Obese Patients: 60 patients with ASA I-III, of both genders, between 18-75 years of age, with a BMI of 40>30 kg m2 and intubated under general anesthesia
  Interventions: Device: monitoring

INTERVENTIONS:
Device: monitoring — rc02, ORI , spO2

SUMMARY:
The primary aim of this study is to compare the effectiveness of ORI and rcSO2 in predicting hypoxia early in obese patients who are sensitive to hypoxia. Our secondary aim is; To determine whether there is a correlation between the changing trend of ORI and rcSO2 in obese patients.

DETAILED DESCRIPTION:
Standard noninvasive monitoring will be applied to the patients taken to the operating table, and heart rate, mean arterial pressure, peripheral oxygen saturation (SpO2), oxygen reserve index (ORI), regional cerebral oxygen saturation, etCO2 values will be recorded. Cerebral oximeter probe placed in the middle of the forehead (every second Cerebral oxygen saturation will be continuously monitored using a rcSO2 reading) (Massimo)Preoxygenation will be performed until the expiratory O2 concentration is 90% (during spontaneous ventilation, FIO2 will be kept between 100% 6 lt7min flow rate and EtCO2 30-35 mmHg). 2 mg midazolam, 2 ug General anesthesia with /kg fentanyl, 3 mg/kg propofol, 0.6 mg/kg rocuronium and 100% O2 will be applied and intubated with a videolaryngoscope. The breathing circuit will be disconnected from the endotracheal tube until the SpO2 drops to 94%. At that time, the breathing circuit will be connected and the patients will be ventilated with 100% FiO2, 8 ml kg-1 ideal body weight, targeted tidal volume, and 5 cm H2O positive end-expiratory pressure until the ORI plateaus. Throughout this process, ORI and cerebral oxygen saturation will be recorded continuously. ORI and rcO2 data will be compared at seven specific time points ( (1) during the basal period; (2) at the end of preoxygenation when ORI reaches a plateau; (3) at the beginning of intubation; (4) when SpO2 reaches 97%; (5) when SpO2 reaches 94% (6) ORI reaches a plateau again (during ventilation with 100% FiO2), and (7) SpO2 reaches baseline

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* The ages of 18-75
* Obese BMI (40>BMI>30 kgm^2)
* Undergoing intubated elective surgery

Exclusion Criteria:

* Patients with significant cardiopulmonary comorbidities
* BMI>40 kgm^2 and BMI<30 kg m^2
* ASA>3
* Patients under 18 years and over 75 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with ASA I-III, of both genders, between 18-75 years of age, with a BMI of 40>30 kg m2 and intubated under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Oxygen Reserve Index and Regional Cerebral Oxygen Saturation Indetermining Hypoxia in Obese Patients | after intubation time until spO2 reaches to 97% and 94% and ori reaches to the plato.Expected to take approximately five minutes
  The primary aim of this study is to compare the effectiveness of ORI and rcSO2 in predicting hypoxia early in obese patients (BMI 30-40 kg/m^2) (weight and height will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
Comparison of Oxygen Reserve Index and Regional Cerebral Oxygen Saturation Indetermining Hypoxia in Obese Patients | time until spo2 is 94% and 97% and ori reaches to the plato.Expected to take approximately five minutes
  Our secondary aim is; To determine whether there is a correlation between the changing trend of ORI and rcSO2 in obese patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gülten A Arslan, Assos Prof, Principal Investigator — Dr Lütfi Kırdar City Hospital
Locations (1):
- University of Health Science, Kartal Dr Lütfi Kırdar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will share the parameters and results of the study

REFERENCES:
- [Result] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567
- [Result] Fleming NW, Singh A, Lee L, Applegate RL 2nd. Oxygen Reserve Index: Utility as an Early Warning for Desaturation in High-Risk Surgical Patients. Anesth Analg. 2021 Mar 1;132(3):770-776. doi: 10.1213/ANE.0000000000005109. PMID 32815872